CLINICAL TRIAL: NCT00985192
Title: A Phase II Study of the mTOR Inhibitor RAD001 in Previously Treated Patients With Unresectable or Metastatic Adenocarcinoma of the Esophagus and Stomach
Brief Title: Everolimus in Treating Patients With Previously Treated Unresectable or Metastatic Esophageal Cancer or Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000655574; UCLA-TRIO-TORI-GI-06; IRB# 09-07-061-01; NOVARTIS-UCLA-TRIO-TORI-GI-06
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2016-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the esophagus; adenocarcinoma of the stomach; recurrent esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Patients receive oral everolimus once daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: everolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: everolimus
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with previously treated unresectable or metastatic esophageal cancer or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall disease-control rate (complete response, partial response, or stable disease) in patients with previously treated unresectable or metastatic adenocarcinoma of the upper gastrointestinal tract treated with everolimus.

Secondary

* To determine the safety and toxicity of everolimus in these patients.
* To determine the efficacy of everolimus, in terms of time to response, duration of response, time to tumor progression, progression-free survival, and overall survival, in these patients.
* To explore potential correlations between clinical outcome and biomarkers of interest, including S6 protein overexpression and/or other mTOR-related proteins in blood and tumor biopsy samples from these patients.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Blood, serum, and tumor tissue samples are collected for biomarker analysis.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of adenocarcinoma of the upper gastrointestinal tract
* Metastatic or unresectable disease
* Received 1-2 prior chemotherapy or biological therapy regimens for unresectable or metastatic disease
* Measurable disease in ≥ 1 dimension by CT scan or MRI
* Patients whose only measurable lesion is a metastatic lymph node are eligible provided they have permission from the principal investigator
* ECOG performance status 0-1
* Life expectancy > 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5.0 times ULN if there is liver metastasis)
* Creatinine clearance > 60 mL/min
* Fasting serum cholesterol < 300 mg/dL or < 7.75 mmol/L*
* Fasting triglycerides < 2.5 times ULN*
* INR ≤ 3.5 (for patients on warfarin)
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 4 months after completion of study treatment (oral, implantable, or injectable contraceptives are not considered effective contraception for this study)
* More than 30 days since prior chemotherapy, surgery, radiotherapy, or investigational agents

Exclusion Criteria:

* uncontrolled diabetes mellitus, defined as fasting serum glucose > 1.5 times ULN
* severely impaired lung function
* known HV infection
* active, bleeding diathesis
* unstable angina pectoris, symptomatic congestive heart failure, or myocardial infarction within the past 6 months
* serious uncontrolled cardiac arrhythmia
* active or uncontrolled infection requiring parenteral antimicrobials
* known liver disease (e.g., cirrhosis, chronic active hepatitis, or chronic persistent hepatitis)
* inability to swallow, impaired gastrointestinal (GI) function, or GI disease (e.g., ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) that would significantly alter the absorption of study drugs or preclude the use of oral medications
* other malignancy within the past 5 years except for nonmelanoma skin cancer or cervical carcinoma in situ
* known hypersensitivity to everolimus, sirolimus, or temsirolimus or to their excipients
* other medical conditions that, in the opinion of the investigator, would preclude study participation
* prior mTOR inhibitors (e.g., rapamycin, CCI-779)
* concurrent chronic treatment with steroids or another immunosuppressive agent
* concurrent prophylactic use of hematopoietic growth factors
* concurrent anticancer agents or therapy (including radiotherapy)
* other concurrent experimental agents
* concurrent strong inhibitors or inducers of the isoenzyme CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev A. Wainberg, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (18):
- United States (18):
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Jude Heritage Medical Group at Virginia K. Crosson Cancer Center, Fullerton, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Pacific Shores Medical Group, Long Beach, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Translational Oncology Research International (TORI) Network, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - TORI REDONDO BEACH (Cancer Care Associates Medical Group, Inc.), Redondo Beach, California
  - Sansum Medical Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Trivalley Oncology Hematology, Westlake Village, California
  - Suburban Hematology-Oncology Associates, P.A., Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 49 patients were enrolled between December of 2007 and November of 2009 from 18 participating sites including the University of California Los Angeles hospitals and clinics participating in the TRIO-US Network.
Groups:
- Everolimus: Patients receive oral everolimus once daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity
  everolimus
  laboratory biomarker analysis
Period: Overall Study
Arm/Group | Everolimus
Started | 49
Completed | 45
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 1
Not completed — Determined to be Ineligible During Trial | 2

BASELINE CHARACTERISTICS:
Population: Of the 49 subjects enrolled, only 45 were determined to be evaluable due to subject withdrawal, an adverse event, and 2 subjects later determined to be ineligible. 45 is the analysis population
Arm/Group | Everolimus
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 64 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 37
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28
  Hispanic | 10
  Asian | 4
  Black | 3
Region of Enrollment [Number; unit: participants]
  United States | 45
Disease Site [Number; unit: participants]
  Gastric | 21
  Gastroesophageal Junction | 13
  Esophagus | 11
Eastern Cooperative Oncology Group (ECOG) score [Number; unit: participants] — The ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. Evaluation is made during examination by a Physician.
  0 - Asymptomatic 1 - Symptomatic but completely ambulatory 2 - Symptomatic, <50% in bed during the day 3 - Symptomatic, >50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours) 4 - Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair) 5 - Death
  participants
    0 | 15
    1 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease-control Rate in Patients With Previously Treated Unresectable or Metastatic Adenocarcinoma of the Upper Gastrointestinal Tract Treated With Everolimus.
Description: Disease control rate (DCR), defined as complete response (CR) + partial response (PR) + stable disease (SD) according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
Time Frame: Radiologic disease assessment was performed every 8 weeks (14 days = 1 cycle) treatment discontinuation.
Measure: Number (95% Confidence Interval); unit: percent subjects with disease control
Arm/Group | Everolimus
Number analyzed (Participants) | 45
percent subjects with disease control | 40 [23 to 54.8]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS), defined as the time from date of initial treatment to date of death. Survival function was estimated using the Kaplan-Meier method.
Time Frame: 2.5 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 45
months | 3.4 [2.7 to 5.6]

3. Secondary Outcome: Efficacy in Terms of Progression Free Response
Description: Progression-free survival (PFS), was defined as the time from the date of initial treatment to first objective documentation of disease progression, or death. Estimated using the Kaplan-Meier method. Complete response (CR) + partial response (PR) + stable disease (SD) were determined according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Radiologic disease assessments were utilized.
Time Frame: evry 3 months in year 1, every 6 months after that
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 45
months | 1.8 [1.7 to 2.2]

4. Secondary Outcome: Observed Biomarkers
Description: Potential correlations between clinical outcome and biomarkers of interest, including S6 protein overexpression and/or other mTOR-related proteins in tumor tissue samples from these patients.
Time Frame: 30 months
Population: Exploratory analysis of translational endpoints in patient samples, Representative paraffin blocks were required for all participating patients. Tissue blocks were obtained on 39 patients.
  p-s6 and p-mTOR IHC expression in tumors
Measure: Number; unit: number of tissue blocks
Arm/Group | Everolimus
Number analyzed (Participants) | 39
number of tissue blocks
  Tumor Grade 0, p-S6 | 4
  Tumor Grade 1+, p-S6 | 15
  Tumor Grade 2+, p-S6 | 8
  Tumor Grade 3+, p-S6 | 9
  Tumor Grade 4+, p-S6 | 3
  Tumor Grade 0, p-mTOR | 0
  Tumor Grade 1+, p-mTOR | 8
  Tumor Grade 2+, p-mTOR | 22
  Tumor Grade 3+, p-mTOR | 9
  Tumor Grade 4+, p-mTOR | 0

5. Secondary Outcome: Biomarker Correlations: Progression Free Survival
Description: Potential correlations between progression free survival and S6 protein and mTOR-related proteins in tumor tissue samples from these patients.
Time Frame: 30 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 39
months
  p-S6 level 0-2 | 1.8 [1.6 to 1.9]
  p-S6 level >2 | 3.5 [1.9 to 3.9]
  p-mTOR level 0-2 | 1.8 [1.6 to 2.1]
  p-mTOR level >2 | 2.6 [.7 to 3.9]

6. Secondary Outcome: Biomarker Correlations: Time to Progression
Description: Potential correlations between time to progression and S6 protein and mTOR-related proteins in tumor tissue samples from these patients.
Time Frame: 30 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 39
months
  p-S6 level 0-2 | 1.75 [1.6 to 1.8]
  p-S6 level >2 | 3.4 [1.9 to 3.9]
  p-mTOR level 0-2 | 1.8 [1.6 to 2.1]
  p-mTOR level >2 | 2.6 [.7 to 3.9]

ADVERSE EVENTS:
Time Frame: Adverse Event data collected continuously for subjects. Subjects evaluated every 14 days until 30 days after last drug dose. Up to 2.5 years.
Description: Systemic adverse event assessment occurred every 14 days through investigator assessment during Treatment.
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 24/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=47)
Mucositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Fatigue (General disorders) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=47)
Alkaline phosphatase (Skin and subcutaneous tissue disorders) | 3 (3)
ALT (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 17 (31)
Anorexia (Metabolism and nutrition disorders) | 14 (18)
AST (Hepatobiliary disorders) | 4 (4)
Bloating (General disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cachexia (General disorders) | 1 (1)
Cardiac Infarction (Cardiac disorders) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dehydration (General disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Distension (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 2 (2)
Dry Mouth (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Dysphagia (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Edema - limb (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 22 (39)
Fever (Infections and infestations) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Halitosis (General disorders) | 1 (1)
Hemorrhage pulmonary - nose (Surgical and medical procedures) | 4 (4)
Hemorrhage, GI - abdomen NOS (Vascular disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Hypercholesteremia (Blood and lymphatic system disorders) | 9 (10)
Hyperglycemia (Blood and lymphatic system disorders) | 7 (13)
Hyperlipidemia (Blood and lymphatic system disorders) | 1 (1)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 5 (5)
Hypocalcemia (Blood and lymphatic system disorders) | 2 (3)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection - Kidney (Infections and infestations) | 1 (1)
Infection - Lung (Infections and infestations) | 1 (1)
Infection - urinary tract NOS (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 1 (1)
LDL - elevated (Blood and lymphatic system disorders) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 3 (5)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Mood alteration - anxiety (Psychiatric disorders) | 1 (1)
Mood alteration - depression (Psychiatric disorders) | 1 (1)
Mucositis - oral cavity (Musculoskeletal and connective tissue disorders) | 11 (17)
Muscle weakness - generalized (General disorders) | 1 (1)
Nasal/paranasal reactions (Ear and labyrinth disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 13 (15)
Neuropathy-sensory (Nervous system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 5 (7)
Pain - abdomen (Nervous system disorders) | 8 (11)
Pain - back (Nervous system disorders) | 1 (1)
Pain - body (Nervous system disorders) | 1 (1)
Pain - chest/thorax NOS (Nervous system disorders) | 1 (1)
Pain - extremity-limb (Nervous system disorders) | 1 (1)
Pain - eye (Nervous system disorders) | 1 (1)
Pain - head (Nervous system disorders) | 2 (2)
Pain - hip (Nervous system disorders) | 1 (1)
Pain - NOS (Nervous system disorders) | 1 (1)
Pain - oral cavity (Nervous system disorders) | 1 (1)
Pain - shoulder (Nervous system disorders) | 1 (1)
Pain - Stomach (Gastrointestinal disorders) | 1 (1)
Pain - throat (Nervous system disorders) | 2 (2)
Performance status decrease (General disorders) | 6 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 11 (17)
Stomatitis (Ear and labyrinth disorders) | 2 (3)
Sweating (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Taste alteration (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (39)
Vomiting (Gastrointestinal disorders) | 8 (10)
Weakness (General disorders) | 2 (2)
Weight loss (General disorders) | 3 (4)

LIMITATIONS AND CAVEATS:
This study had several limitations with the major weakness being that it was a single- rm, non-comparative study. At the time this study was launched, a Japanese report indicating a DCR was 50 % was not yet reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No